CLINICAL TRIAL: NCT05081596
Title: PATH-Pain: A Primary Care-Based Psychosocial Intervention To Improve Cognitive and Depression Outcomes in Older Adults With MCI and Early Stage AD
Brief Title: A Primary Care-Based Psychosocial Intervention To Improve Cognitive & Depression Outcomes in Older Adults With MCI & Early Stage AD
Acronym: PATH-Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-01023108; R01AG070055 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Depression; Pain; Cognitive Impairment
Keywords: Older Adults; Mild Cognitive Impairment; Early Stage Alzheimer's Disease
MeSH Terms: conditions — Depression; Pain; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem Adaptation Therapy for Pain (PATH-Pain) (Experimental): Problem Adaptation Therapy-PAIN (PATH-PAIN) is an emotion regulation intervention aimes to reduce stress and decrease depression and disability.
  Interventions: Behavioral: PATH-Pain
- Attention Control Usual Care (No Intervention): Usual Care involves the continued medical attention and treatment provided by the subject's physician and other medical professionals in primary care. This may include medical intervention or referrals to specialists to address issues of depression, pain or memory difficulties. Subjects will also be asked to meet with a study research assistant for structured interviews and educational sessions consisting of general questions regarding health habits and other non-medical topics unrelated to cognitive impairment, pain, and depression. Additionally, subjects will receive an educational booklet on pain and depression.

INTERVENTIONS:
Behavioral: PATH-Pain — The goals of PATH-Pain are to: 1) Teach problem solving skills to reduce negative emotions, by using emotion regulation and problem- solving strategies to overcome these difficulties. 2) Use compensatory strategies and environmental adaptation tools (notes, checklists, calendars, etc.) to avoid limitations resulting from memory problems, help improve emotion regulation, and create an easier environment to live in. If found helpful and participant agrees, a tablet application called WellPATH will be used to help the subject with emotion regulation techniques. The tablet will be given at the beginning of treatment and will be returned at the end of treatment. 3) Invite caregiver participation, when appropriate.
  Subjects in the PATH-PAIN group will receive 8 weekly sessions (first 8 weeks) with a study therapist and 6 monthly phone sessions (3 individual and 3 group) for 9-36 weeks. Each session will last approximately 50 minutes.
  Arms: Problem Adaptation Therapy for Pain (PATH-Pain)

SUMMARY:
The purpose of the study is to examine the effect of Problem Adaptation Therapy for Pain (PATH-Pain) on cognitive functioning, depression and pain-related disability in 100 older adults with cognitive impairment, chronic pain, and depression. The study will test if PATH-Pain has better cognitive, affective, and functional outcomes than Attention Control Usual Care.

DETAILED DESCRIPTION:
This is a Randomized Control Trial to target cognition in older adults with MCI or Early AD, depression, and chronic pain with a psychotherapeutic intervention in primary care. This project will study the efficacy of 8 in-office acute treatment sessions (first 8 weeks) and 6 telephone delivered sessions (3 individual and 3 group) in the following months (from 9-36 weeks) of PATH- Pain vs. an equal number of sessions consisting of Attention Control Usual Care in improving cognitive, affective, and functional outcomes. Each therapy session will last approximately 50 minutes. Assessments will be conducted at study entry and weeks 5, 9 (end of acute treatment; includes assessment of cognitive functioning), 24, 36 (end of follow-up treatment; includes assessment of cognitive functioning) and 52 (includes assessments of cognitive functioning) after randomization. This is an efficacy trial, but by being delivered by certified mental health clinicians, it has a strong "real-world" focus.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* MCI or early stage probable or possible AD diagnosis (as defined by Albert et al or McKhann et al) al). Patients will have at least mild cognitive deficits defined by 16 ≤ MoCA ≤ 25.
* Montgomery Asberg Depression Rating Scale (MADRS)[55] total ≥ 5, which reflects at least some mild depressive symptoms.
* Participants will be off antidepressants, cholinesterase inhibitors or memantine or on a stable dosage for at least 12 weeks.
* Chronic pain (neuropathic, nociceptive or mixed disorders): presence of pain on most days for at least 3 months and average pain intensity score >=4.
* Clinical Dementia Rating 0.5 ≤ (CDR) ≤ 1.
* Participant will have capacity to consent.
* Participation of a study partner (e.g. caregiver/family member/significant other) is required.

Exclusion Criteria:

* Deemed to have a significant suicide risk as assessed by site PI and clinical team.
* Deemed too unstable medically or neurologically to safely enroll in a research trial.
* Deemed too psychiatrically unstable to safely enroll in randomized trial of psychotherapy.
* Requiring psychiatric hospitalization at baseline for safety.
* Lack of English fluency.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive functioning, as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, Weeks 9, 36, 52
  RBANS is a widely used neuropsychological instrument which assesses cognitive functioning. The lowest score is 40 (severe cognitive impairment) and highest is 160 (less cognitive impairment).

SECONDARY OUTCOMES:
Change in cognition, as measured by the Alzheimer's Disease Assessment Scale - Cognition Subscale (ADAS-COG) | Baseline, Weeks 9, 36, 52
  ADAS-Cog is a widely used measure of cognition in clinical trials for antidementia therapies. The lowest score is 0 (no cognitive impairment) and highest is 70 (severe cognitive impairment).
Change in depressive symptoms, as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, Weeks 5, 9, 24, 36, 52
  MADRS is a depression instrument that has been used in studies of older adults with and without cognitive deficits. The lowest score is 0 (no depressive symptoms) and highest score is 60 (severe depressive symptoms).
Change in pain-related disability, as measured by the Roland-Morris Scale | Baseline, Weeks 5, 9, 24, 36, 52
  Roland-Morris is a widely used instrument which measures pain-related disability. The lowest score is 0 (no disability) and highest score is 24 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University; Mannigton C Reid, MD, Principal Investigator — Weill Medical College of Cornell University; Lisa Ravdin, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: http://nda.nih.gov/